CLINICAL TRIAL: NCT06942312
Title: Elucidating Hepatic Metabolism in Non-alcoholic Fatty Liver Disease
Acronym: ECHO
Status: Enrolling by invitation | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Luukkonen, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: HUS/176/2025
Record Dates: First submitted 2025-03-14; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Hepatic mitochondrial dysfunction; Non-alcoholic Fatty Liver Disease NAFLD; 13C-α-Ketoisocaproic Acid Breath Test; liver stiffness
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, breath samples, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Advanced NAFLD: Intrahepatic triglyceride content ≥ 5.56 % as determined by magnetic resonance specroscopy and liver stiffness measurement ≥ 8 kPa using transient elastography (Fibroscan)
  Interventions: Diagnostic Test: Ketoisocaproic acid breath test; Diagnostic Test: Ammonium Chloride; Diagnostic Test: Bicarbonate de sodium; Diagnostic Test: Deuterated Water; Diagnostic Test: Oral Glucose Tolerance Test
- Mild NAFLD: Intrahepatic triglyceride content ≥ 5.56 % as determined by magnetic resonance specroscopy and liver stiffness measurement < 8 kPa using transient elastography (Fibroscan)
  Interventions: Diagnostic Test: Ketoisocaproic acid breath test; Diagnostic Test: Ammonium Chloride; Diagnostic Test: Bicarbonate de sodium; Diagnostic Test: Deuterated Water; Diagnostic Test: Oral Glucose Tolerance Test
- Healthy control: Intrahepatic triglyceride content < 5.56 % as determined by magnetic resonance specroscopy and liver stiffness measurement < 8 kPa using transient elastography (Fibroscan)
  Interventions: Diagnostic Test: Ketoisocaproic acid breath test; Diagnostic Test: Ammonium Chloride; Diagnostic Test: Bicarbonate de sodium; Diagnostic Test: Deuterated Water; Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Ketoisocaproic acid breath test — 13C-alpha-ketoisocaproic acid breath test to estimate hepatic mitochondrial reductive stress (1 mg/kg body weight; oral dose; study duration 390 min)
Diagnostic Test: Ammonium Chloride — 15N-ammonium chloride stable isotope test to estimate ureagenesis (20 mg/kg body weight; oral dose; study duration 390 min)
Diagnostic Test: Bicarbonate de sodium — 13C-bicarbonate breath test to estimate body bicarbonate pool size and gastric emptying (0.5 mg/kg body weight; oral dose; study duration 390 min)
Diagnostic Test: Deuterated Water — Deuterated water stable isotope test to estimate hepatic de novo lipogenesis and gluconeogenesis (3 g/kg body water; oral dose; duration: overnight)
Diagnostic Test: Oral Glucose Tolerance Test — A standard 2-hour 75-gram oral glucose tolerance test to assess glucose tolerance and whole body metabolism

SUMMARY:
The goal of this observational, cross-sectional, case-control clinical study is to investigate the metabolic adaptations underlying the progression of nonalcoholic fatty liver disease (NAFLD), and to test the hypothesis that hepatic mitochondrial reductive stress contributes to progression of NAFLD.

The main question it aims to answer is:

Do patients with advanced NAFLD compared to patients with mild NAFLD and healthy controls have increased hepatic mitochondrial reductive stress as determined by the ketoisocaproate breath test and by plasma beta-hydroxybutyrate to acetoacetate ratio (b-OHB/AcAc)?

DETAILED DESCRIPTION:
In this study the investigators study the metabolic adaptations underlying the progression of nonalcoholic fatty liver disease (NAFLD), namely hepatic mitochondrial reductive stress, ureagenesis, de novo lipogenesis and gluconeogenesis in patients with advanced and mild NAFLD and in healthy controls.

At the first visit, an informed consent will be obtained, followed by assessment of inclusion/exclusion criteria and medical history. Participants fulfilling the criteria will be enrolled in the study. A physical examination will be performed and laboratory test will be taken. Body composition will be determined with bioelectrical impedance and dual-energy x-ray absorptiometry (DEXA).

At the second visit, hepatic lipid content will be measured with magnetic resonance spectroscopy.

At the third visit, participants will pick up containers for overnight urine collection and doses of deuterated water and a standardized meal replacement bar. The fourth visit is a clinical study visit. In a specified order, participants will drink tracer doses of 15NH4Cl, 13C-bicarbonate and 13C-alpha-ketoisocaproate. An oral glucose tolerance test is performed in the end of the study day. Breath samples are collected at different time points for determination of 13C enrichment of CO2. Furthermore, "arterialized" blood samples are taken to obtain beta-hydroxybutyrate to acetoacetate ratios (b-OHB/AcAc) at different timepoints.

Whole-body oxidation of lipids, carbohydrates and protein will be determined using indirect calorimetry.

ELIGIBILITY:
The following inclusion/ exclusion criteria will be employed:

1. Participants must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subject must be likely to be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge.
3. Participants must be aged between 18-75 years.
4. Participants are not allowed to have alcohol consumption of 350 g/week or more in women and 420 g/week or more in men.
5. Participants are not allowed to have history of liver disease other than NAFLD as judged by history and physical examination and standard laboratory tests.
6. Participants are not allowed to have claustrophobia or metal implants to allow magnetic resonance studies.
7. Participants are not allowed to be pregnant or lactating.
8. No known or anticipated difficulties in cannulation of peripheral veins.
9. No history or evidence of any other clinically significant disorder, condition or disease other than those outlined above that, in the opinion of the investigator may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety, or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population and hospital outpatients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic mitochondrial reductive stress as determined by plasma beta-hydroxybutyrate-to-acetoacetate ratio | Fourth study visit (2 months)
  Ratio of beta-hydroxybutyrate and acetoacetate concentrations in arterialized plasma
Hepatic mitochondrial reductive stress as determined by the ketoisocaproic acid breath test | Fourth study visit (2 months)
  Breath 13CO2 enrichment after ingesting 13C-alpha-ketoisocaproate measured as area under the curve

SECONDARY OUTCOMES:
Plasma metabolomics | Fourth study visit (2 months)
  Arterialized plasma analyzed by nuclear magnetic resonance
Plasma metabolomics | Fourth study visit (2 months)
  Arterialized plasma analyzed by mass spectrometry

OTHER OUTCOMES:
Fractional Rate of Ureagenesis | Fourth study visit (2 months)
  Hepatic incorporation of ammonia to urea (i.e. ureagenesis), as determined by plasma [15N1]urea enrichment after ingestion of a tracer dose of 15NH4Cl
Fractional Rate of Hepatic de novo lipogenesis | Fourth study visit (2 months)
  Hepatic de novo lipogenesis, as determined by deuterium enrichment in plasma triglyceride-palmitate after ingestion of tracer doses of deuterated water
Fractional Rate of Gluconeogenesis | Fourth study visit (2 months)
  Fractional gluconeogenesis, as determined by deuterium enrichment in plasma glucose after ingestion of tracer doses of deuterated water
Ammonia incorporation to glutamine | Fourth study visit (2 months)
  Hepatic incorporation of ammonia to glutamine (i.e. glutamine synthesis), as determined by plasma [15N1]glutamine enrichment after ingestion of a tracer dose of 15NH4Cl
Bicarbonate pool size | Fourth study visit (2 months)
  Breath 13CO2 enrichment after ingesting 13C-bicarbonate measured as area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Panu K. Luukkonen, MD, PhD, Principal Investigator — University of Helsinki
Locations (1):
- Helsinki Central University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to European Union GDPR regulations.